CLINICAL TRIAL: NCT00153764
Title: Effectiveness of a One-a-Day Cooper Complete Vitamin / Mineral Supplement With or Without Omega-3 Fatty Acid Ingestion
Brief Title: Effectiveness of a Vitamin Mineral Supplement
Acronym: Omega-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cooper Institute (Other)
Collaborators: Cooper Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CI0039
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: supplement; omega-3 fatty acid; Homocysteine; LDL cholesterol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- multivitamin (Placebo Comparator): 1 tablet morning and evening
  Interventions: Drug: Cooper Complete One-A-Day Vitamin Supplement

INTERVENTIONS:
Drug: Cooper Complete One-A-Day Vitamin Supplement

SUMMARY:
The goal of the study is to evaluate the effectiveness of a new one-a-day Cooper complete vitamin supplement with or without a combined omega-3 fatty acid supplement on selected clinical risk factor measures. Participants taking the Cooper Complete one-a-day vitamin plus omega-3 fatty acid will have greater improvement in homocysteine, LDL cholesterol, and C-reactive protein than those taking the other supplements.

DETAILED DESCRIPTION:
Participants will be randomized to 1 of 3 groups: vitamin with omega-3, vitamin w/o omega-3, or omega-3 alone. They will take the vitamin 12 weeks, after which time they will return for all laboratory tests. Persons who are currently taking a supplement must undergo a 2-week washout period before beginning the study. Participants taking the Cooper Complete one-a-day vitamin plus omega-3 fatty acid will have greater improvement in homocysteine, LDL cholesterol, and C-reactive protein than those taking the other supplements.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years of age, maintain current diet and exercise regimen, not currently taking vitamins or agree to stop for 6 weeks

Exclusion Criteria:

* BMI <18.5 or >34.9, recent blood donation, elevated blood pressure, cholesterol, or fasting blood glucose that requires medication, plans to move soon, or pregnant or plans to become pregnant

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
homocycsteine
LDL cholesterol oxidation rate

SECONDARY OUTCOMES:
fasting plasma glucose
C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Conrad Earnest, PhD, Principal Investigator — The Cooper Institute
Locations (1):
- The Cooper Institute, Dallas, Texas, United States